CLINICAL TRIAL: NCT01842139
Title: Randomized Phase I Study Combining Suppression of T Regulatory Cells With WT1 Vaccine Therapy for AML Patients in Complete Remission
Brief Title: Vaccine Therapy and Basiliximab in Treating Patients With Acute Myeloid Leukemia in Complete Remission
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0545; NCI-2011-03588 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-03; First posted 2013-04-29 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22)
MeSH Terms: conditions — Congenital Abnormalities | interventions — Basiliximab; montanide ISA 51; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (vaccine with Montanide) (Experimental): Patients receive WT1 126-134 peptide vaccine emulsified in Montanide ISA 51 VG SC on day 0 and then once every 2 weeks.
  Interventions: Biological: WT1 126-134 peptide vaccine; Drug: Montanide ISA 51 VG; Other: laboratory biomarker analysis
- Arm B (vaccine with poly-ICLC) (Experimental): Patients receive WT1 126-134 peptide vaccine in poly-ICLC SC on day 0 and then once every 2 weeks.
  Interventions: Biological: WT1 126-134 peptide vaccine; Drug: poly ICLC; Other: laboratory biomarker analysis
- Arm C (vaccine therapy, monoclonal antibody) (Experimental): Patients assigned to Arm C receive basiliximab IV over 30 minutes on day -7 and WT1 126-134 peptide vaccine as in Arm A or Arm B, whichever had a superior cellular immune response.
  Interventions: Biological: basiliximab; Biological: WT1 126-134 peptide vaccine; Drug: Montanide ISA 51 VG; Drug: poly ICLC; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: basiliximab — Given IV
  Other Names: SDZ-CHI-621; Simulect
  Arms: Arm C (vaccine therapy, monoclonal antibody)
Biological: WT1 126-134 peptide vaccine — Given SC
Drug: Montanide ISA 51 VG — Given SC
  Arms: Arm A (vaccine with Montanide); Arm C (vaccine therapy, monoclonal antibody)
Drug: poly ICLC — Given SC
  Other Names: Hiltonol; poly I:poly C with poly-1-lysine stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; stabilized polyriboinosinic/polyribocytidylic acid
  Arms: Arm B (vaccine with poly-ICLC); Arm C (vaccine therapy, monoclonal antibody)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I trial studies the side effects and best way to give vaccine therapy together with basiliximab in treating patients with acute myeloid leukemia (AML) in complete remission. Vaccines made from the WT1 peptide may help the body build an effective immune response to kill cancer cells. Montanide ISA 51 VG and poly-ICLC may enhance this response. Monoclonal antibodies, such as basiliximab, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether WT1 126-134 peptide vaccine with Montanide ISA 51 VG is more effective than with poly-ICLC when given together with basiliximab in treating AML

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the immunogenicity of WT1 peptide (WT1 126-134 peptide vaccine) emulsified in Montanide (Montanide ISA 51 VG) in elderly patients with AML.

II. To determine whether toll-like receptor 3 (TLR3) agonist (poly-L-lysine and carboxymethyl cellulose [poly ICLC]) could be a potent immunologic adjuvant, and increases the frequencies of WT1-specific T cells following vaccination.

III. To determine whether depletion of regulatory T cells occurs upon administration of the anti-cluster of differentiation (CD)25 monoclonal antibody Basiliximab, and whether this is associated with increased frequencies of WT1-specific T cells following vaccination.

IV. To assess whether WT1 vaccination +/- TLR3 agonist (poly ICLC) combined with Basiliximab results in decreased levels of WT1 transcripts in peripheral blood cells compared to WT1 vaccination +/- TLR3 as measured by quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR).

SECONDARY OBJECTIVES:

I. To examine the safety and gain preliminary information on efficacy of WT1 peptide vaccination +/- TLR3 agonist (poly ICLC) combined with Basiliximab.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive WT1 126-134 peptide vaccine emulsified in Montanide ISA 51 VG subcutaneously (SC) on day 0 and then once every 2 weeks.

ARM B: Patients receive WT1 126-134 peptide vaccine emulsified in poly-ICLC SC on day 0 and then once every 2 weeks.

ARM C: Patients assigned to Arm C receive basiliximab intravenously (IV) over 30 minutes on day -7 and WT1 126-134 peptide vaccine as in Arm A or Arm B, whichever had a superior cellular immune response.

In all arms, treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients may then receive 6 additional monthly vaccinations.

After completion of study treatment, patients are followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Hematological malignancies, including AML, MDS, CML in blast phase and other conditions at the investigator's discretion.
* Bone marrow biopsy-confirmed CR or CRi, more than CR1 is allowed, such as CR2 or CR3. The enrollee is deemed not a candidate for stem cell transplant due to advanced age or co-morbidities; or the enrollee does not have donor available; or enrollee refuses stem cell transplant due to personal belief; or stem cell transplant is not current standard of care. Patients who are post stem cell transplant in CR or CRi are allowed if they are off immunosuppression,and not treated with systematic steroid for GVHD
* Karnofsky performance status index > or = 80%
* Written informed consent
* Absolute neutrophil count > or = 500/μl
* Platelet count >= 20,000/μl with transfusion
* Creatinine = or < 2 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) = or < 5 x ULN
* Bilirubin = or < 3 x ULN
* Human leukocyte antigens (HLA) typing: patient must express HLA-A2
* Age > 18 years and < 85 years
* Electrocardiogram (EKG) without evidence of arrhythmia or changes that indicate acute ischemia
* Pulse oximetry showing oxygen saturation of at least 90% on room air
* No irreversible coagulopathy, international normalized ratio (INR) =< 2
* No sign of tumor lysis syndrome, uric acid needs to be in normal range prior to treatment
* Not in diabetic ketoacidosis (DKA), sickle cell crisis, and not having severe peripheral vascular disease on active anti-coagulation treatment

Exclusion Criteria:

* Pregnant or nursing women; women who still have child-bearing potential must be tested for urinary or serum beta human chorionic gonadotropin (βHCG)
* Biological or chemotherapy in the 4 weeks prior to the start of dosing
* Patients with intrinsic immunosuppression, including seropositivity for human immunodeficiency virus (HIV) antibody; patients should be tested for HIV
* Serious concurrent infection, including active tuberculosis, hepatitis B, or hepatitis C; patients should be tested for hepatitis B surface antigen and hepatitis C antibody; patients who are hepatitis C antibody (Ab) positive can be eligible if they are PCR negative
* Active or history of confirmed autoimmune disease
* Concurrent systemic corticosteroids (except physiologic replacement doses) or other immunosuppressive drugs (eg. cyclosporin A)
* Active or history of autoimmune disease including but not limited to rheumatoid arthritis (rheumatoid factor [RF]-positive with current or recent flare), inflammatory bowel disease, systemic lupus erythematosus (clinical evidence with antinuclear antibody [ANA] 1:80 or greater), ankylosing spondylitis, scleroderma, multiple sclerosis, autoimmune hemolytic anemia, and immune thrombocytopenic purpura; seropositivity alone will not be considered positive
* Psychiatric illness that may make compliance to the clinical protocol unmanageable or may compromise the ability of the patient to give informed consent; patients with clinical evidence of dementia should have a competent designee participate in decision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-12-05 (Actual); Primary Completion 2015-02-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Comparison of peptide specific immunologic response between regimens | Over 9 months
  Evaluated by flow cytometry and using IFN-gamma ELISPOT as the primary measures. Compared using a two-sample t test.
Comparison of regulatory T cells (Treg) number changes between regimens | 9 months
  Evaluated by flow cytometry and using interferon (IFN)-gamma Enzyme-linked immunosorbent spot (ELISPOT) as the primary measures. Compared using a two-sample test. The Treg cell counts and percentage by flow cytometry, the FoxP3 expression by qRT-PCR, and the peptide specific CD8+cell level by ELISPOT will be measured continuously prior to basiliximab and WT1 126-134 peptide vaccine and after basiliximab and/or WT! 126-134 peptide vaccine.

SECONDARY OUTCOMES:
Molecular response in terms of WT1 expression | Every 12 weeks for 1 year after stopping treatment
Relapse-free survival | Every 12 weeks for 1 year after stopping treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Liu, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Liu H, Zha Y, Choudhury N, Malnassy G, Fulton N, Green M, Park JH, Nakamura Y, Larson RA, Salazar AM, Odenike O, Gajewski TF, Stock W. WT1 peptide vaccine in Montanide in contrast to poly ICLC, is able to induce WT1-specific immune response with TCR clonal enrichment in myeloid leukemia. Exp Hematol Oncol. 2018 Jan 11;7:1. doi: 10.1186/s40164-018-0093-x. eCollection 2018. PMID 29344432